CLINICAL TRIAL: NCT05324306
Title: Extremity Occlusion With Tourniquets Increases Proximal Systolic Pressure
Brief Title: Tourniquets Increase Proximal Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 00109291
Record Dates: First submitted 2022-04-04; First posted 2022-04-12 (Actual); Results first posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Blood Pressure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Application of Tourniquets on Lower Extremities (Experimental): Participants will have their baseline blood pressure measured in their upper extremities followed by application of CAT tourniquets to both lower extremities. Blood pressure will be measured again in the upper extremities once the CAT tourniquets are deployed. This will be repeated 3 times.
  Interventions: Device: combat application tourniquets (CAT)

INTERVENTIONS:
Device: combat application tourniquets (CAT) — CAT tourniquets have been indicated for use in emergency situations revolving around a wounded limb, such as hemorrhage control.22-23 CAT tourniquets are the official tourniquet of the US Army since in 2005.
  We will deploy well-studied and FDA approved combat application tourniquets (CAT) on both thighs of volunteer healthy adult subjects while measuring blood pressure in the upper extremities.

SUMMARY:
There is an urgent clinical need to improve survival and neurologic outcomes after cardiac arrest. When a patient goes into cardiac arrest, cardiopulmonary resuscitation (CPR) with chest compressions is the current standard of care treatment to mechanically circulate blood through the patient's body. The immediate and long-term success of CPR is critically dependent on the maintenance of adequate coronary and cerebral perfusion. The investigators propose that CPR outcomes can be improved by capitalizing on the innate mechanism of vasoconstriction and preferentially routing the limited oxygenated blood to the heart and brain. The proposed solution is occlusion of extremity vasculature will increase coronary and cerebral perfusion and improve patient outcomes after cardiac arrest. Prior research has investigated the efficacy of manipulating peripheral vascular resistance with tourniquets in animal studies with improved cardiac and cerebral perfusion and survival. To prove this is an adequate solution in humans, the investigators plan to use tourniquets on the legs to occlude the peripheral vasculature in healthy humans and measure more proximal blood pressure before and after tourniquet deployment. Proof of concept of this solution will make way for development of novel devices for use during cardiac arrest and CPR to improve heart and brain perfusion and ultimately improve cardiac arrest outcomes.

The investigators will recruit 30 healthy human participants and measure their blood pressure in their arm. They will then place two commercially-available, FDA-approved tourniquets around each thigh to stop blood flow to the legs. The investigators will measure the blood pressure in the arms again. They will then release the tourniquets after blood pressure measurement. This will be repeated three times with breaks between each repetition.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults with no known chronic medical conditions between the ages of 18 and 60 years old willing and able to consent themselves.
* Subjects who are native English speakers or self-report as fluent in English.

Exclusion Criteria:

* Subjects who have a history of or are a current smoker, have a history of or current illicit drug use, have a history of or current alcohol abuse.
* Subjects who self-report as pregnant.
* Subjects who self-report diabetes, cardiac disease including hypertension requiring medication, or a history of compartment syndrome or peripheral vascular disease.
* Subjects with known chronic diseases not listed above, including but not limited to Rheumatoid Arthritis, McArdle's disease, etc.
* Subjects with elevated blood pressure (>130/80mmHg) on the day of the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-08-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seigler SW, Quinn KM, Holman HL, Kim JY, Rajab TK. A single-center, nonblinded, clinical trial comparing blood pressures before and after tourniquet application in healthy humans: A study protocol. PLoS One. 2023 Jan 6;18(1):e0280139. doi: 10.1371/journal.pone.0280139. eCollection 2023. PMID 36608001

RESULTS

PARTICIPANT FLOW:
Groups:
- Application of Tourniquets on Lower Extremities: Participants will have their baseline blood pressure measured in their upper extremities followed by application of CAT tourniquets to both lower extremities. Blood pressure will be measured again in the upper extremities once the CAT tourniquets are deployed. This will be repeated 3 times.
  combat application tourniquets (CAT): CAT tourniquets have been indicated for use in emergency situations revolving around a wounded limb, such as hemorrhage control.22-23 CAT tourniquets are the official tourniquet of the US Army since in 2005.
  We will deploy well-studied and FDA approved combat application tourniquets (CAT) on both thighs of volunteer healthy adult subjects while measuring blood pressure in the upper extremities.
Period: Overall Study
Arm/Group | Application of Tourniquets on Lower Extremities
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Application of Tourniquets on Lower Extremities
Number analyzed (Participants) | 27
Age, Continuous [Mean (Full Range); unit: years] | 25.74 [22 to 35]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 27
Systolic Blood Pressure [Mean (Full Range); unit: mmHg] | 122 [115 to 129]
Diastolic Blood Pressure [Mean (Full Range); unit: mmHg] | 72 [65 to 81]
Heart Rate [Mean (Full Range); unit: bpm] | 70 [57 to 83]

OUTCOME MEASURES:

1. Primary Outcome: Systolic Blood Pressure During Application of the CAT Tourniquets
Description: We define the primary study endpoint as successful application of CAT tourniquets in normal physiology in healthy humans with a minimum increase in blood pressure of 10 mmHg measured in the arms.
Time Frame: the average of 3 repetitions is reported; the duration of each tourniquet application was 5 minutes and participants rested 3-5 minutes between each repetition
Measure: Mean (Full Range); unit: mmHg
Arm/Group | Application of Tourniquets on Lower Extremities
Number analyzed (Participants) | 27
mmHg
  Systolic Blood Pressure | 129 [120 to 138]
  Diastolic Blood Pressure | 76 [69 to 83]

ADVERSE EVENTS:
Time Frame: Up to 1 year
Arm/Group | Application of Tourniquets on Lower Extremities
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2022-11-10): https://cdn.clinicaltrials.gov/large-docs/06/NCT05324306/Prot_000.pdf